CLINICAL TRIAL: NCT04221633
Title: R34 Family Navigator E3 Project: Enhance Early Engagement in Mental Health Services Through Children's Advocacy Center's Family Advocates
Brief Title: R34 Family Navigator Enhancing Early Engagement
Acronym: NavE3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 11290; R34MH118486 (NIH)
Record Dates: First submitted 2019-12-13; First posted 2020-01-09 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Mental Health Issue; Trauma, Psychological
MeSH Terms: conditions — Psychological Trauma | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: The current clinical trial involves three conditions (N=25 each): webinar-training only, webinar training plus consultation, and waitlist control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Webinar only (Experimental): Participants in this arm will attend a webinar training program (3 webinars over the course of 4 to 8 weeks) to receive training in evidence-based engagement strategies, trauma, evidence-based practices, and mental health screening.
  Interventions: Behavioral: Enhancing Early Engagement (E3) webinar
- Webinar plus consultation (Experimental): Participants in this arm will receive the same webinar training as subjects in arm 1, but they will also receive 10 consultation calls over the course of four months to further develop their skills in engaging families and screening for mental health services.
  Interventions: Behavioral: Enhancing Early Engagement (E3) webinar; Behavioral: Consultation for E3 training
- Delayed training group (No Intervention): This group will not receive any training for the duration of the study year, in order to serve as a waitlist control group. They will be eligible to receive the training after the randomized control trial has been completed.

INTERVENTIONS:
Behavioral: Enhancing Early Engagement (E3) webinar — Webinar-based training to provide information regarding evidence-based engagement strategies (e.g., motivational interviewing, McKay's engagement model), trauma, mental health screening, and identifying evidence-based mental health treatments for children.
  Arms: Webinar only; Webinar plus consultation
Behavioral: Consultation for E3 training — 10 consultation calls with experts in engagement, child trauma, and mental health screening to support the webinar training
  Arms: Webinar plus consultation

SUMMARY:
For the current study, the investigators will develop, implement, and evaluate web-based and consultative training for Family Advocates employed at Children's Advocacy Centers (CACs) across the United States to enhance children's early engagement in evidence-based mental health treatment. The interactive web-based training will embed key targets of knowledge and skills related to family engagement, trauma, evidence-based practices (EBP), and EBP services in the community. Seventy-five CACs who apply to participate in training will be randomized to a webinar-only training group, a webinar plus consultation training group, and a delayed (waitlist) control group. It is hypothesized that the Family Advocates and CAC Directors will report high levels of satisfaction with the training. More importantly, it is also hypothesized that webinar training will improve Family Advocates' knowledge, resulting in minor improvement in EBP engagement, while the addition of consultation in the second training group will lead to increased use of engagement skills, thereby resulting in greater improvement in family engagement in EBP.

DETAILED DESCRIPTION:
Partnering with the accrediting board for CACs, the National Children's Alliance (NCA), the investigators will implement and evaluate training for Family Advocates to enhance early engagement in EBP (E3 training). Two levels of E3 training will be tested. The first level, webinar-only (E3w), will be web-based training on MH screening, EBP identification, trauma and effects of trauma, and engagement strategies that directly target known hindrances to accessing EBP in high risk, traumatized populations. The second level, webinar plus consultation (E3w+c), will add short-term consultation with experts in engagement and mental health. Consultation will target Family Advocates' skills in engagement, mental health screening, and coordination of care through strategies found to enhance skill acquisition. The investigators propose to test two key mechanisms of change for improving EBP engagement: knowledge (e.g., EBP identification) and skills (e.g., addressing caregiver perceptions of MH). To examine these change mechanisms, the investigators will implement the feasibility study designed to accomplish three tasks: (1) test if E3w training provides incremental benefits in engagement rates over the no training comparison group, (2) examine if E3w+c further improves outcomes beyond the E3w engagement rates and (3) examine mediating and moderating factors impacting outcome and implementation, including cost. The hypotheses that E3w will improve Family Advocates' knowledge, resulting in minor improvement in EBP engagement, and that addition of consultation in E3w+c will lead to increased use of engagement skills, resulting in greater improvement in family engagement in EBP, will be tested.

Using NCA's innovative data capture systems, including the Outcome Management System (OMS; designed to obtain follow-up surveys from families and multidisciplinary team members), as well as a specific data tracking procedure using REDCap, the investigators will track case management details (including mental health needs and referrals) from each site randomized. In addition, knowledge learned via the training (pre- and post-knowledge assessments) will be tracked. In addition, NCA quantitative data on family engagement in EBP will be drawn, and the data submitted and integrated with pre- and post-training surveys of Family Advocates and CAC leaders measuring knowledge and perceptions of the training, including its utility, strengths, weaknesses, and costs.

Applications were released to CACs nationwide in October of 2019, and sites were officially selected and randomized to groups using an adaptive randomization procedure such that a broad range of the selected covariates that are hypothesized to influence key outcomes occurs in all conditions. Participants from sites, including Advocates and Senior Leaders, will officially consent and enroll in the study in mid-December 2019. Participants will provide study data via an online data platform (i.e., REDCap). The outcomes of interest are the time-varying and CAC-varying provider fidelity and knowledge, as well as the family screening and engagement in treatment. Linear mixed effects models will be used to evaluate these outcomes, with generalized versions of these applied whenever the distribution of the outcome variable and the residuals suggest these to be appropriate

ELIGIBILITY:
Inclusion Criteria:

* Fully accredited by NCA
* Directly provides EBP for child mental health or has established and demonstrated linkages for services in the community
* Participates in OMS
* Has Memorandum of Understanding (MOU) or data sharing agreements with all referral sources
* Both CAC directors and Family Advocate(s) must demonstrate commitment to the training and data collection procedures.

Exclusion Criteria:

* There are no specific exclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Rate of child engagement in mental health services | Tracked over the course of one year for all families seen at the CAC.
  Caregiver report (via Outcome Management System [OMS] survey on a yes/no item) if family attended the first appointment of mental health services they were referred to be the CAC.
Score on 45-item Knowledge Assessment | Through study completion, up to one year
  Questionnaire of knowledge-based multiple choice and true/false questions, assessing knowledge of evidence-based engagement skills, trauma, evidence-based treatments, and mental health screening, yielding a total correct out of 45
Rate of evidence-based Engagement Skills survey | Through study completion, up to one year
  Advocate self-report of use of evidence-based engagement skills via a 39-item survey with skills utilized ranked on 5-point Likert scale (not at all to extensively); Caregiver report of advocate use of skills via three items on the OMS Survey, rating Advocate use of skills on a 4-point Likert scale (strongly agree to Strongly Disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Jane F Silovsky, Ph.D., Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - National Children's Alliance, Washington D.C., District of Columbia
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided
Currently working with NIMH to determining data archiving process.

REFERENCES:
- [Derived] Taylor EK, Dopp AR, Lounsbury K, Thompson Y, Miller M, Jorgensen A, Silovsky JF. Enhancing Early Engagement (E3) in mental health services training for children's advocacy center's victim advocates: feasibility protocol for a randomized controlled trial. Pilot Feasibility Stud. 2021 Dec 6;7(1):212. doi: 10.1186/s40814-021-00949-2. PMID 34872619